CLINICAL TRIAL: NCT03369379
Title: Randomized, Double-blind, Placebo-controlled Trial to Measure the Efficacy and Safety of Vitamin D3 in Patients With Fibromyalgia.
Brief Title: Valuation of Efficacy and Safety of Vitamin D3 Use in 80 Women Diagnosed With Fibromyalgia. Using FIQ Score and VAS.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Luis Ivan Lozano Plata, Dr., Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RE16-00019
Record Dates: First submitted 2017-07-27; First posted 2017-12-12 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Fibromyalgia; D Vitamin Deficiency
Keywords: Fibromyalgia; D Vitamin
MeSH Terms: conditions — Fibromyalgia; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Longitudinal, prospective, interventional, randomized.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind, the subject of study and researcher.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- D3 Vitamin (Active Comparator): In this group subjects will receive 1 vitamin D3 capsule of 50,000 units, each week, for 12 weeks.
  Interventions: Drug: D3 Vitamin
- Placebo (Placebo Comparator): In this group the subjects will receive 1 placebo capsule each week for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: D3 Vitamin — Subjects will receive a capsule of 50,000 units of vitamin D3 echa week for 12 weeks, basal levels of vitamin D will be taken and again at week 12.
  Other Names: D3
  Arms: D3 Vitamin
Other: Placebo — Placebo pill
  Arms: Placebo

SUMMARY:
Fibromyalgia is a disease that significantly decreases the quality of life of people who suffer from it, has great repercussions at the socio-economic level due to the incapacity it produces. It is characterized by generalized pain, fatigue, sleep disorders, psychological stress and mental alterations, besides presenting painful points in different parts of the body to physical examination. Having few effective treatments is necessary to explore new options in their management to improve the general conditions of the patient. Previous studies have shown that patients with fibromyalgia have had low levels of vitamin D in the blood, a favorable response from post-vitamin D supplementation has been seen. This vitamin has been associated with pain pathways and with increased The perception of the same when it is in smaller amount. We will select patients with Fibromyalgia diagnosis from the external consultation of Rheumatology of the University Hospital "Dr. José Eleuterio González "of the UANL, over 18 years old who have not been previously supplemented with vitamin D, will initially be measured in blood of vitamin D, in addition to calcium as a safety measure, we will have a group that will only receive placebo and Another that will be supplemented with 50 thousand units weekly for 12 weeks, we will apply a questionnaire that measures pain scale and another one that measures the impact of the disease in the daily life of the patient, this will be done in a beginning and at the end of the 12 weeks .

DETAILED DESCRIPTION:
Fibromyalgia is a disease characterized mainly by generalized pain, with great repercussion in the patient's quality of life as well as in his work and social performance. There are different therapies that have not been totally effective for the management of this pathology, for that reason it is necessary to look for cost-effective options and the reach of all the patients to obtain remission of the symptoms.

Fibromyalgia affects 1-4% of the general population, patients manifest chronic pain and other comorbidities such as sleep disorders, fatigue, depression, psychological stress and cognitive disturbances. It is a significant cause of loss of employment and disconnection from the social environment.

A longitudinal, prospective, randomized study with patients diagnosed with Fibromyalgia will be performed at the outpatient clinic of the Rheumatology Service at the University Hospital "Dr. José Eleuterio González "of the Autonomous University of Nuevo León.

DEFINITION OF VARIABLES

Dependent variable:

Vitamin D levels Conceptual definition: it is considered as pro-hormone, its active metabolite 1-25-dihydroxyvitamin D functions as a hormone since it has its own receptors found in all human cells.4 Operational definition: Normal levels> 30-100 ng / ml, 10-30 ng / ml insufficiency and a deficit <10 ng / ml as defined by the laboratory.19 Measurement scale: qualitative.

Independent variables:

Fibromyalgia Impact Questionnaire (FIQ) Conceptual definition: a questionnaire that assesses the impact of FM in physical capacity, the possibility of doing the usual work and, in the case of performing a paid work, the degree to which FM has affected this activity as well As subjective items very related to the FM picture (pain, fatigue, tiredness and stiffness) and emotional state (anxiety and depression).

Operational definition: consists of three domains functionality, global impact and symptomatology. It consists of 10 items. The first is the only one containing several sub-items (a-j), in number of 10, each with a rank of 4 points (from 0, always, to 3, never) according to a Likert scale.

This item evaluates the functional capacity of the patient through questions about activities related to daily life: buy, drive, etc. The second and third items correspond to numerical scales that refer to days of the week: the second on a scale from 1 to 7, and the third from 1 to 5. The rest of the items are valued using analog visual scales (EVA) From 0 to 10.

Type of variable: Quantitative dichotomous.

Visual Analogue Scale (VAS) Conceptual definition: approach used to measure pain. In one line the patient scores a point that best describes the intensity of his pain.

Operational definition: a scale that allows to measure the intensity of pain, draws a line that divides from 0 to 10, on the left corresponds to the use of pain with the number 0, on the right is the maximum degree of pain corresponds to 10 .

Type of variable: quantitative

Other variables:

Age Conceptual definition: Time that has lived a person counting since birth. Operational definition: Age expressed in years according to the clinical file. Type of variable: quantitative.

Gender Conceptual definition: set of people or things that has common general characteristics.

Operational definition: male and female according to the clinical file. Type of variable: Qualitative.

C-reactive protein (CRP) Conceptual definition: plasma protein or acute phase reactant that rises during inflammatory processes.

Operational definition: it was considered elevated when its levels exceeded 1 mg / dl as it marks the laboratory. It was taken as positive or negative according to this commented level.

Erythrocyte sedimentation rate (ESR) Conceptual definition: acute phase reactant, measures the time it takes erythrocytes to fall or decant in a period of time. It is elevated in inflammatory, infectious and neoplastic processes.

Operational definition: elevated ESR levels were considered according to the formula adjusted for age in men = age / 2, for women = age + 10/2.

MEASUREMENT TOOLS

Fibromyalgia Impact Questionnaire (FIQ) Questionnaire that measures the impact that Fibromialgia has on the daily life of the patient. It is responsible for evaluating three items: functionality of the subject, overall impact of the disease and symptomatology. It was developed in 1980 by Drs. Carol Burckhardt, Sharon Clark and Robert Bennett Portland, Oregon USA. Published 1991, revisions 1997 - 2002 - 2009. It is one of the most used tools for evaluation of patients with FM. It consists of 10 items. The first is the only one containing several sub-items (a-j), in number of 10, each with a rank of 4 points (from 0, always, to 3, never) according to a Likert scale. This item evaluates the functional capacity of the patient through questions about activities related to daily life: buy, drive, etc. The second and third items correspond to numerical scales that refer to days of the week: the second on a scale from 1 to 7, and the third from 1 to 5. The rest of the items are valued using visual analogue scale (VAS) From 0 to 10. It was validated by Monterde in 2004.

Visual Analog Scale (VAS) Scale that allows to measure the intensity of pain, draws a line that divides from 0 to 10, on the left corresponds to the use of pain with the number 0, on the right is the maximum degree of pain corresponds to 10.

Mini Neuro-Psychiatric Interview It is a brief and highly structured interview of the major psychiatric disorders of ICD-10 and DSM-IV. It was elaborated by Y. Lecrubier et al. Of the "Salpétrére" of Paris and D. Scheehan et al. Of the University of Tampa Florida in 1992, 1994 and 1998. It serves to diagnose depressions, phobias, suicides, generalized anxiety disorders, agoraphobia, substance abuse or dependence. A tool of great utility in primary care.

SAMPLE SIZE:

According to Young's nomogram for sample size calculation for controlled clinical trials (with an alpha of 0.05 and statistical power of 0.8), the sample size (including a 20% to compensate for possible losses) by study group is : 80 patients.

SAMPLING TECHNIQUE:

Patients were selected using a non-probabilistic sampling technique for consecutive cases.

STATISTIC ANALYSIS:

The t-test for independent samples and logistic regression will be used to evaluate the effect of the independent variables on the dependent variable. A value of p ≤ 0.05 shall be considered significant. The statistical package SPSS version 17.0 for Windows 7 will be used.

METHODS Allocation method: Consecutive incident patients will be included, those eligible for the study will be assigned to treatment groups using a pre-established allocation table, which was generated in the randomization module of the True Epistat statistical program.

DESCRIPTION OF THE STUDY

1. Four visits are planned for the evaluation of subjects.
2. At the first visit, the subjects attend the consultation 12 of the Department of Rheumatology at the University Hospital "Dr. José Eleuterio González "where they are evaluated by a rheumatologist to confirm the diagnosis of Fibromyalgia according to the criteria of the American College of Rheumatology of 1990 and 2010. The Fibromyalgia Impact Questionnaire (FIQ) will be applied at baseline and the Visual Analog Scale (VAS).
3. Once the diagnosis of Fibromyalgia has been made, at the same first visit, a joint ultrasound will be performed by Rheumatologist expert in the field, in order to evaluate the presence of synovitis only in those patients with Primary Fibromyalgia.
4. All patients included in the Fibromyalgia Diagnostic Study will continue with their standard established treatment for the disease and may receive salvage treatment for pain management if they so require.
5. On the second visit, 15 ml of blood sample will be taken through venipuncture. 4ml of serum will be stored in aliquots of 0.5mL each in a freezer at -80 ° C located in the laboratory of the Rheumatology Service, in order to determine basal levels of vitamin D. Levels of c-reactive protein and Sedimentation to correlate them with the clinical data of inflammation obtained to the interrogation. We will determine levels of serum calcium to rule out the possibility of hypercalcemia at the start of the study and as a safety measure. In the case of clinical suspicion of Fibromyalgia secondary to rheumatoid arthritis, the study of rheumatoid factor and anti-cyclic citrullinated peptide antibodies will be carried out. The Mini-Neuro-psychiatric Interview will be applied by an expert Psychiatrist from the UANL, previously trained to perform this task.
6. At the second visit, subjects will be randomized to placebo or 50,000 international units of Vitamin D3 weekly for 12 weeks. It should be noted that neither the Rheumatologist who performed the Fibromyalgia diagnosis nor the person who will be responsible for providing the placebo or the vitamin will know the contents of the capsules. A double-blind study is planned.
7. At week 6 of the study a telephone call will be made to all patients to assess adverse effects.
8. The third visit will be performed at week 12 of the study, subjects from both groups are again assessed through the FibromyalgiaImpact Questionnaire (FIQ) and Visual Analogue Scale (VAS). A 15 ml blood sample will be taken to determine vitamin D levels as well as serum calcium levels for monitoring adverse effects.
9. After completing 12 weeks of vitamin D supplementation or placebo as appropriate. All subjects in the placebo group will have the option of receiving vitamin D3 supplementation 50,000 IU orally in capsules per week for 12 weeks and then on a fourth visit they will be given a 15ml blood sample to measure vitamin D levels. It means that the study will be opened to know the subjects who received placebo after having completed the first twelve weeks. The blood samples obtained will be stored in the Laboratory of the Department of Rheumatology only during the duration of the study.

DATA COLLECTION SYSTEM A patient file will be included (Case report form). Finally, the data will be transferred to the database and analyzed with the SPSS program for Windows 7 version 17.0.

ELIGIBILITY:
Inclusion Criteria:

* Female patients older than 18 years.
* Patients who agree to participate in the study.
* Those that meet the ACR 1990 and 2010 criteria for Fibromyalgia.
* No previous use of vitamin D.
* Patients diagnosed with primary or secondary fibromyalgia.

Exclusion Criteria:

* Those subjects with previous use of vitamin D.
* Known subjects with renal, liver, calcium metabolism disorders, malabsorption disorders, known neoplasms.
* Subjects with serum calcium levels equal to or greater than 10.2 mg / dl.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women diagnosed with Fibromyalgia from the outpatient clinic of the "Dr. José Eleuterio González" University Hospital of the Autonomous University of Nuevo Leon.
Enrollment: 80 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
FIBROMYALGIA IMPACT QUESTIONNAIRE | 12 weeks
  Number of items in scale: The version from 19911 consisted of 10 items with 10 sub-items in the physical function scale (total items + sub-items = 19). The modified version from 1997 consists of 20 items with 11 physical function items (total items + sub-items = 30). The 2009 version consists of 21 items across the 3 domains of Function (n = 9), Overall Impact (n = 2), and Symptoms (n = 10).
  Subscales: Subscales from the 1991 version1 include physical function (10 sub-items), feel good (1 item), missed work (1 item), do job (1 item), pain (1 item), fatigue (1 item), rested (1 item), stiffness (1 item), anxiety (1 item), and depression (1 item).

SECONDARY OUTCOMES:
VISUAL ANALOGUE SCALE | 12 weeks
  Visual analogue scales (VAS) are psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients and use this to achieve a rapid (statistically measurable and reproducible) classification of symptom severity and disease control.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Alberto Garza Elizondo, Ph D, Principal Investigator — Hospital Universitario "Dr. José Eleuterio González"
Locations (1):
- Universidad Autónoma de Nuevo León, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Yes
It will be agreed with all participating researchers.
Supporting Information: SAP, CSR
Time Frame: 5 years
Access Criteria: On request

REFERENCES:
- [Background] Yong WC, Sanguankeo A, Upala S. Effect of vitamin D supplementation in chronic widespread pain: a systematic review and meta-analysis. Clin Rheumatol. 2017 Dec;36(12):2825-2833. doi: 10.1007/s10067-017-3754-y. Epub 2017 Aug 15. PMID 28812209